CLINICAL TRIAL: NCT02128386
Title: A Study on Medication Adherence and "True" Resistance in Patients Referred to a Medical Outpatient Department in Germany With the Diagnosis "Resistant Hypertension".
Brief Title: Medication Adherence and "True" Resistance in Patients With Resistant Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Jürgen Scholze, Head of the Medical Outpatient Department of the Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: EA1/328/13
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Hypertensive Disease; Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for therapeutic drug monitoring
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Renal sympathetic denervation: Olmesartan 40 mg once daily + Amlodipine 5 or 10 mg once daily + Hydrochlorothiazide 25 mg one daily plus renal sympathetic denervation
- Intensified antihypertensive treatment: Olmesartan 40 mg once daily + Amlodipine 5 or 10 mg once daily + Hydrochlorothiazide 25 mg one daily plus second-line antihypertensive agents (e.g. mineralocorticoid receptor antagonists or alpha-1-blockers)

SUMMARY:
The purpose of this study is to estimate the proportion of patients with "true" resistance among patients referred to the Medical Outpatient Department of the Charité - Universitätsmedizin Berlin with the diagnosis "resistant hypertension". Moreover, data on medication adherence will be collected based on therapeutic drug monitoring and on the answers to validated questionnaires. Finally, efficacy, safety and costs of renal sympathetic denervation will be compared to an intensified drug treatment in an exploratory way.

ELIGIBILITY:
Inclusion Criteria:

* Female or male adult patients with arterial hypertension and admission diagnosis of "resistant hypertension"
* Informed consent
* Exclusion of secondary arterial hypertension
* Kidney function (estimated glomerular filtration rate [eGFR] ≥ 45 ml/min/1.73 m2)

Exclusion Criteria:

* Age < 18 years
* Secondary arterial hypertension
* Type 1 Diabetes mellitus
* Unstable coronary heart disease, myocardial infarction or stroke in the last 6 months
* Psychiatric diseases
* Significant carotid stenosis (> 70%)
* Pregnancy
* Chronic kidney disease (eGFR < 45 ml/min/1.73 m2)
* Severe liver injury (elevation of transaminases more than twofold the upper limit of normal)
* Abuse of alcohol or illegal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female patients referred to the Medical Outpatient Department of the Charité - Universitätsmedizin Berlin with the diagnosis "Resistant hypertension".
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Estimation of the proportion of patients with "true" resistance among patients referred to the Medical Outpatient Department of the Charité - Universitätsmedizin Berlin with the diagnosis "resistant hypertension" | Week 6

SECONDARY OUTCOMES:
Assessment of all costs of both treatments within one year. | During the whole course of the study (24 weeks) and for another 24 weeks after the end of the study
Analysis of medication adherence at baseline, after fixed-dose triple combination treatment and in the end of the study via therapeutic drug monitoring, and correlation of these results with the questionnaire findings. | Baseline, week 6, end of study on week 24
Explorative evaluation of the efficacy of renal sympathetic denervation compared to an intensified drug treatment based on ambulatory blood pressure and ambulatory blood pressure measurement over 24 hours. | Week 6 - week 24
Assessment of adverse events in order to evaluate the safety of both treatments. | During the whole course of the study (24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Scholze, Professor, Principal Investigator — Charite - Universitätsmedizin Berlin; Reinhold Kreutz, Professor, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Medical Outpatient Department of the Charité - Universitätsmedizin Berlin, Berlin, Germany